CLINICAL TRIAL: NCT03200132
Title: Respiratory Motion Correction of Cardiac Combined Positron Emission Tomography and Magnetic Resonance Imaging (PET/MRI)
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-4-156
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac PET/MRI — For patients undergoing 18-Fluor- fluorodeoxyglucose (18F-FDG) PET/MRI or PET/Computed Tomography (CT), additional cardiac PET/MRI scans are acquired.

SUMMARY:
This study evaluates the possibility of Magnetic Resonance Imaging (MRI) based respiratory motion correction of simultaneously acquired cardiac Positron Emission Tomography (PET) images.

ELIGIBILITY:
Inclusion Criteria:

* 18F-FDG injection for clinical diagnostic PET/MRI or PET/CT

Exclusion Criteria:

* Diet-suppressed myocardial uptake of 18F-FDG
* General exclusion criteria for MRI (i.e. metallic implants, claustrophobia, pregnancy, etc.)
* Not willing to be informed about incidental findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving 18F-FDG for clinical diagnostic PET/MRI or PET/CT.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Target-to-background ratio (TBR) | 15-20 minutes

SECONDARY OUTCOMES:
Signal-to-noise ratio (SNR) | 15-20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wildberger, MD PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands